CLINICAL TRIAL: NCT02465346
Title: "Mobile Stroke Unit"-Concept for Delivery of Specialized Acute Stroke Care to Patients in Remote Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: USaarland
Record Dates: First submitted 2015-05-31; First posted 2015-06-08 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Acute Stroke
Keywords: acute stroke; prehospital; treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSU-based stroke management (Experimental): The Mobile Stroke Unit (MSU) and the conventional emergency medical Service (EMS) will meet at the emergency site. The patient's medical history, the physical examination will directly be performed by a physician. Laboratory tests will be analyzed by a point of care laboratory. CT will be performed. After performance of the acute stroke diagnostic work-up the patients and, if indicated thrombolysis, the patient will be transported according to the diagnostic results: Stroke due to large vessel occlusion or to intracranial hemorrhage-> Neurovascular centre; Stroke without large vessel occlusion or without hemorrhage-> primary hospital with regional stroke unit.
  Interventions: Device: MSU-based stroke management
- Control stroke management (Active Comparator): After performing patient's medical history, physical examination (reassessment of the extended Face Arm Speech Time score) and glucose testing by the (stroke trained) emergency personnel, the patient will be transported according to current best clinical practice and relevant guidelines to the next stroke unit or neurovascular centre. The hospital stroke team will be prenotified by the EMS. According to the patients needs the patient might be further transferred.
  Interventions: Device: Control stroke management

INTERVENTIONS:
Device: MSU-based stroke management — Prehospital stroke treatment with a mobile stroke unit
  Arms: MSU-based stroke management
Device: Control stroke management — Conventional stroke management
  Arms: Control stroke management

SUMMARY:
Treatment of acute stroke must be fast. The aim of this trial is to show feasibility, safety and clinical benefit of a strategy of diagnosis and treatment directly at the emergency site for hyperacute treatment and transfer to the most appropriate target hospital. The effects on reduction delays until different stroke treatments will be assessed. First estimations of cost-effectiveness will also be performed.

DETAILED DESCRIPTION:
Stroke is a medical emergency for which "time-is-brain". Indeed, a huge body of animal experimental and clinical evidence exists that demonstrates that reducing the time to thrombolytic therapy is the most important variable in prevention of the disability. However, most stroke patients arrive to hospital too late for any type of acute stroke treatment: Only an estimated 19-60% of stroke patients present within 3 hours after symptom onset. Today, for stroke patients 3 different treatment options exist.

1. Thrombolysis with recombinant tissue plasminogen activator (rt-PA) is an effective treatment for many acute stroke patients as evidenced by several large randomized trials.
2. More recently, mechanical clot removal via catheters has been developed. There is currently increasing evidence that in obstruction of large brain vessels such endovascular treatment is superior to systemic thrombolysis in regard to recanalization rates and outcome.
3. Patients with intracranial hemorrhage can profit if transferred to hospitals with neurosurgical treatment options such as ventricular drainage or hematoma removal.

However, each of these treatment are highly time sensitive and due the availability of endovascular and neurosurgical treatment options only in very few highly specialized neurovascular centres decision in which institution the patient should be transported is of high medical and financial relevance. The aim of this trial is to show feasibility, safety and clinical benefit of a strategy of diagnosis and treatment directly at the emergency site and its role in decision regarding transfer to appropriate target institution, thus potentially allowing reduction of time until treatment and delays until specialized treatment also in remote regions. First estimations of cost-effectiveness will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of acute stroke reported to the EMS dispatcher office (extended FAST Score, Table I) and verified by the EMS (after glucose testing)
* Reported onset of symptoms until call ≤ 8 hours
* Patients with "wake up stroke"
* Age older than 18 years
* Patient (or representative) is willing to participate voluntarily and to sign a written informed consent.

Exclusion Criteria:

* Cardiopulmonary unstable medical conditions requiring immediate treatment in an intensive care unit
* Patients with preexisting severe functional impairment and disease
* Known allergy or contraindications to contrast agents

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Proportion of stroke patients with accurate decision regarding transfer to the most appropriate target hospital | within 3 month

SECONDARY OUTCOMES:
Proportion of patients with large vessel occlusion a) being directly transferred to a neurovascular centre, and b) being evaluated/ treated by an interventionalist | within 3 month
Time between symptom onset/alarm and evaluation/treatment by an interventional radiologist in case of large vessel occlusion | within 3 month
Proportion of patients with haemorrhage being a) directly transferred to a neurovascular centre, and being b) evaluated/treated by a neurosurgeon. | within 3 month
Time between symptom onset/alarm and evaluation/treatment by a neurosurgeon in case of haemorrhage | within 3 month
Proportion of patients treated with rt-PA and time between symptom onset/ alarm and start of thrombolysis | within 3 month
Functional neurological status (mRS) (D7, D90) | within 3 month
Proportion of secondary transfers of stroke patients between primary stroke unit and neurovascular centre in all stroke patients, and in subgroups with ischemic and hemorrhagic stroke | within 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Klaus C Fassbender, MD, Principal Investigator — Department of Neurology, Saarland University
Locations (1):
- Department of Neurology, University Hospital of the Saarland, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Result] Walter S, Kostopoulos P, Haass A, Keller I, Lesmeister M, Schlechtriemen T, Roth C, Papanagiotou P, Grunwald I, Schumacher H, Helwig S, Viera J, Korner H, Alexandrou M, Yilmaz U, Ziegler K, Schmidt K, Dabew R, Kubulus D, Liu Y, Volk T, Kronfeld K, Ruckes C, Bertsch T, Reith W, Fassbender K. Diagnosis and treatment of patients with stroke in a mobile stroke unit versus in hospital: a randomised controlled trial. Lancet Neurol. 2012 May;11(5):397-404. doi: 10.1016/S1474-4422(12)70057-1. Epub 2012 Apr 11. PMID 22497929
- [Derived] Helwig SA, Ragoschke-Schumm A, Schwindling L, Kettner M, Roumia S, Kulikovski J, Keller I, Manitz M, Martens D, Grun D, Walter S, Lesmeister M, Ewen K, Brand J, Fousse M, Kauffmann J, Zimmer VC, Mathur S, Bertsch T, Guldner J, Magull-Seltenreich A, Binder A, Spuntrup E, Chatzikonstantinou A, Adam O, Kronfeld K, Liu Y, Ruckes C, Schumacher H, Grunwald IQ, Yilmaz U, Schlechtriemen T, Reith W, Fassbender K. Prehospital Stroke Management Optimized by Use of Clinical Scoring vs Mobile Stroke Unit for Triage of Patients With Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Dec 1;76(12):1484-1492. doi: 10.1001/jamaneurol.2019.2829. PMID 31479116